CLINICAL TRIAL: NCT06280703
Title: A Four-Part, Randomized, Double-Blind (Part A) and Open-Label (Part B, Part C, and Part D), Multi-Dose, Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3938577 in Healthy Participants and Participants With Type 1 Diabetes Mellitus
Brief Title: A Study of LY3938577 in Healthy Participants and Participants With Type 1 Diabetes Mellitus (T1DM)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 18792; J4P-MC-IYAB (Other: Eli Lilly and Company); U1111-1301-8386 (Other: Universal Trial Number); 2023-510365-10-00 (Other: EU Trial Number)
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Lispro

STUDY DESIGN:
Intervention Model Description: Crossover Assignment Parallel (Part A) and Crossover design (Part B, Part C, and Part D)
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator) Double-Blind (Part A) and Open-Label (Part B, Part C, and Part D)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (10):
- Part A Period 1: LY3938577 (Experimental): Single dose of LY3938577 administered intravenously (IV) in healthy participants.
  Interventions: Drug: LY3938577
- Part A Period 1: Placebo (Placebo Comparator): Single dose of Placebo administered intravenously (IV) in healthy participants.
  Interventions: Drug: Placebo
- Part B: LY3938577 (Experimental): For each euglycemic and hyperglycemic clamps participants with T1DM will receive single doses of LY3938577 administered intravenously with Insulin Lispro administered at a constant low rate to cover individual participant's basal (fasting) insulin demand to maintain a stable glucose level.
  Interventions: Drug: LY3938577; Drug: Insulin Lispro
- Part B: Insulin Degludec (Active Comparator): For each euglycemic and hyperglycemic clamps participants with T1DM will receive single doses of Insulin Degludec administered intravenously with Insulin Lispro administered at a constant low rate to cover individual participant's basal (fasting) insulin demand to maintain a stable glucose level.
  Interventions: Drug: Insulin Degludec; Drug: Insulin Lispro
- Part C: LY3938577 (Experimental): LY3938577 administered subcutaneously (SC)
  Interventions: Drug: LY3938577
- Part C: Insulin Degludec (Active Comparator): Insulin Degludec administered subcutaneously (SC)
  Interventions: Drug: Insulin Degludec
- Part A Period 2: LY3938577 (Experimental): Sequential dose of LY3938577 administered subcutaneously (SC).
  Interventions: Drug: LY3938577
- Part A Period 2: Placebo (Placebo Comparator): Sequential dose of Placebo administered subcutaneously (SC)
  Interventions: Drug: Placebo
- Part D Period 1: Basal Insulin and Lispro Prandial Insulin (Other): Pre-study basal insulin (provided by patient) and lispro prandial insulin administered SC
  Interventions: Drug: Basal Insulin; Drug: Lispro Prandial Insulin
- Part D Period 2: Lispro Prandial Insulin and LY3938577 (Experimental): Lispro prandial insulin and LY3938577 administered SC
  Interventions: Drug: LY3938577; Drug: Lispro Prandial Insulin

INTERVENTIONS:
Drug: LY3938577 — Administered Intravenously (IV)
  Arms: Part A Period 1: LY3938577; Part B: LY3938577
Drug: Placebo — Administered Intravenously (IV)
  Arms: Part A Period 1: Placebo
Drug: Insulin Degludec — Administered Intravenously (IV)
  Arms: Part B: Insulin Degludec
Drug: Insulin Lispro — Administered Intravenously (IV)
  Arms: Part B: Insulin Degludec; Part B: LY3938577
Drug: LY3938577 — Administered subcutaneously (SC)
  Arms: Part A Period 2: LY3938577; Part C: LY3938577; Part D Period 2: Lispro Prandial Insulin and LY3938577
Drug: Placebo — Administered subcutaneously (SC)
  Arms: Part A Period 2: Placebo
Drug: Insulin Degludec — Administered SC
  Arms: Part C: Insulin Degludec
Drug: Basal Insulin — Administered subcutaneously (SC)
  Arms: Part D Period 1: Basal Insulin and Lispro Prandial Insulin
Drug: Lispro Prandial Insulin — Administered subcutaneously (SC)
  Arms: Part D Period 1: Basal Insulin and Lispro Prandial Insulin; Part D Period 2: Lispro Prandial Insulin and LY3938577

SUMMARY:
The main purpose of this study is to look at the amount of the study drug LY3938577 that gets into the blood stream and how long it takes the body to get rid of it. At a later stage of this study (part B and C) the blood sugar lowering effect and the duration of action of LY3938577 will be evaluated compared to Insulin Degludec.

The study will also evaluate the safety and tolerability of LY3938577 and information about any side effects experienced will be collected.

The study will be conducted in four parts (A, B, C, and D). Healthy participants in Part A Period 1 will receive a single dose of LY3938577 or a placebo given via intravenous (IV) infusion. In Part A Period 2, participants will receive a single subcutaneous (SC) dose of either LY3938577 or placebo. Participants in Part B with Type 1 Diabetes Mellitus (T1DM) will receive single doses of either LY3938577 or Insulin Degludec given via IV infusion. Participants in Part C with Type 1 Diabetes Mellitus (T1DM) will receive two doses of either LY3938577 or Insulin Degludec administered SC. Participants in Part D with Type 1 Diabetes Mellitus (T1DM) will be evaluated in 2 periods, with Period 1 administered pre-study basal insulin and lispro mealtime insulin to establish insulin needs, and Period 2 administered lispro mealtime insulin and daily doses of LY3938577.

The study will last up to approximately 11 weeks for Part A, 10 weeks for Part B, 13 weeks for Part C, and 10 weeks for Part D , including screening period.

ELIGIBILITY:
Inclusion Criteria:

Part A -

• Participants who are overtly healthy as determined by medical history and physical examination.

Parts B and C -

* Have Type 1 Diabetes Mellitus (T1DM) for at least 2 years with a fasting C-peptide level of 0.20 Nanomoles Per Liter (nmol/L) or less, or nonfasting C-peptide level of 0.30 nmol/L or less at screening.
* Have well-controlled HbA1c between 6.0% to 8.5 percent (%).
* Insulin pump users with a total daily basal dose between 15 to 45 International Unit (IU).

Part D -

* Have T1DM for at least 1 year with a fasting C-peptide level of 0.20 nmol/L or less, or non-fasting C-peptide level of 0.30 nmol/L or less.
* HbA1c between 6% to 8.5% inclusive.
* Insulin pump users with a total daily basal dose between 15 to 45 International Unit (IU).
* Insulin multiple daily injection users (glargine or degludec insulin) with a total daily insulin dose between 0.3 to <1.2 (I)U/kg/day.
* No hypoglycaemia unawareness.
* Basal insulin dose that is between 30% to 70% of the total daily insulin dose
* Are able to complete the exercise challenge test.

All Parts -

* Have normal blood pressure, pulse rate and safety laboratory test results that are acceptable for the study.
* Have body mass index (BMI) between 18.0 and 35.0 kilograms per meter squared (kg/m²), inclusive, at screening.
* Have venous access sufficient to allow for blood sampling.
* Male and/or female not of childbearing potential.

Exclusion Criteria:

Parts B, C, and D -

* Have had more than 1 emergency room visit or hospitalization due to poor glucose control (hyperglycemia or diabetic ketoacidosis) within the last 6 months prior to screening.
* Have had any episodes of severe hypoglycemia (defined as requiring assistance due to neurologically disabling hypoglycemia), hypoglycemia unawareness, or both within the last 6 months prior to screening.

Parts B and C -

* Have been treated with Glucagon-like Peptide-1 Receptor Agonists (GLP-1 RA), Dipeptidyl Peptidase 4 (DPP4) inhibitor, Glucose-dependent Insulinotropic Polypeptide (GIP) agonists, Metformin, or Sodium-Glucose Transport Protein 2 (SGLT2) inhibitors within the previous 3 months.
* Have received systemic or inhaled glucocorticoid therapy (excluding topical, intraarticular, and intraocular preparations) for more than 14 consecutive days within 4 weeks before screening.

Part D -

• Have been treated with Dipeptidyl peptidase-4 (DPP-IV) inhibitors, GLP-1 RA, GIP/GLP-1 RA, Metformin, Pramlintide, SGLT2 inhibitors, or Neutral Protamine Hagedorn (NPH) insulin within the previous 3 months.

All Parts -

* Have had any of the following cardiovascular conditions: acute myocardial infarction, New York Heart Association Class III or IV heart failure, or cerebrovascular accident (stroke).
* Have gastroparesis or have undergone gastric bypass (bariatric) surgery or restrictive bariatric surgery (for example, Lap-Band®) prior to screening.
* Have history of renal transplantation, currently receiving renal dialysis, have serum creatinine level of more than 2.00 milligrams per decilitre (mg/dL) or have an estimated glomerular filtration rate of less than 60.0 milliliters (mL) / minute /1.73 square meters.
* Have acute or chronic hepatitis, or obvious clinical signs or symptoms of any other liver disease except non-alcoholic fatty liver disease (that is, participants with non-alcoholic fatty liver disease are eligible for participation), and/or have elevated liver enzyme measurements, as determined by the local laboratory at screening and as indicated:

  * Total bilirubin (TBL) >2 × the Upper Limit of Normal (ULN) in the absence of Gilbert's syndrome, or
  * Alanine aminotransferase (ALT) /serum glutamic pyruvic transaminase (SGPT) >2.5 × ULN, or
  * Aspartate aminotransferase (AST) /serum glutamic oxaloacetic transaminase (SGOT) >2.5 × ULN.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Part A: Number of participants with one or more Adverse Event (s) (AEs), and Serious Adverse Event(s) (SAEs) considered by the investigator to be related to study drug administration. | Baseline up to Approximately Week 11
  A summary of AEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module.
Part B and D: Number of participants with one or more Adverse Event (s) (AEs), and Serious Adverse Event(s) (SAEs) considered by the investigator to be related to study drug administration. | Baseline up to Week 10
  A summary of AEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module.
Part A: Number of Participants With Clinically Significant Changes in Vital Signs | Baseline up to Approximately Week 11
Part B: Number of Participants With Clinically Significant Changes in Vital Signs | Baseline up to Week 10
Part A: Number of Participants With Clinically Significant Changes in Safety Laboratory Parameters | Baseline up to Approximately Week 11
Part B: Number of Participants With Clinically Significant Changes in Safety Laboratory Parameters | Baseline up to Week 10
Part A: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3938577 | Predose on day 1 up to week 13 post dose
  PK: AUC of LY3938577 for intravenous administration
Part A: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3938577 | Predose on day 1 up to week 13 post dose
  PK: AUC of LY3938577 for SC administration
Part B: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3938577 | Predose on day 1 up to week 13 post dose
  PK: AUC of LY3938577
Part C: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3938577 | Predose on day 1 up to week 13 post dose
  PK: AUC of LY3938577 for SC administration
Part D: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3938577 | Predose on day 1 up to week 13 post dose
  PK: AUC of LY3938577 for SC administration
Part A: PK: Maximum Observed Concentration (Cmax) of LY3938577 | Predose on day 1 up to week 13 post dose
  PK: Cmax of LY3938577
Part B: PK: Maximum Observed Concentration (Cmax) of LY3938577 | Predose on day 1 up to week 13 post dose
  PK: Cmax of LY3938577
Part C: PK: Concentration of LY3938577 | Predose on day 1 up to week 13 post dose

SECONDARY OUTCOMES:
Part B: Pharmacodynamic (PD): Area under the glucose infusion rate curve (GIR AUC) of LY3938577 | Predose up to day 14 post dose
  Measured at different glucose levels in participants with T1DM
Part C: PD: Glucose infusion rate (GIR) of LY3938577 | Predose up to day 14 post dose
  Measured at different glucose levels in participants with T1DM

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Profil Institut für Stoffwechselforschung, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3938577 in Healthy Participants and Participants With Type 1 Diabetes Mellitus (T1DM) — https://trials.lilly.com/en-US/trial/465015